CLINICAL TRIAL: NCT05302271
Title: Phase IA and IB Study of AAVrh.10hFXN Gene Therapy for the Cardiomyopathy of Friedreich's Ataxia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20-01021274; R61HL151355 (NIH)
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Friedreich Ataxia; Cardiomyopathies; Cardiac Hypertrophy; Myocardial Fibrosis
MeSH Terms: conditions — Friedreich Ataxia; Cardiomyopathies; Cardiomegaly | interventions — Prednisone

STUDY DESIGN:
Intervention Model Description: The clinical study design is a dose-escalation study with 4 cohorts of n=25, 5 subjects at each of 3 doses to establish the safety of the investigational drug product, and 1 cohort with n=10 at the maximum tolerated dose. The vector will be delivered intravenously.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- First Dose Cohort (Experimental): AAVrh.10hFXN will be administered intravenously.
  Interventions: Biological: AAVrh.10hFXN, serotype rh.10 adeno-associated virus (AAV) gene transfer vector expressing the cDNA coding for human FXN; Drug: Prednisone
- Second Dose Cohort (Experimental): AAVrh.10hFXN will be administered intravenously.
  Interventions: Biological: AAVrh.10hFXN, serotype rh.10 adeno-associated virus (AAV) gene transfer vector expressing the cDNA coding for human FXN; Drug: Prednisone
- Third Dose Cohort (Experimental): AAVrh.10hFXN will be administered intravenously.
  Interventions: Biological: AAVrh.10hFXN, serotype rh.10 adeno-associated virus (AAV) gene transfer vector expressing the cDNA coding for human FXN; Drug: Prednisone
- Maximum Tolerated Dose Cohort (Experimental): AAVrh.10hFXN will be administered intravenously.
  Interventions: Biological: AAVrh.10hFXN, serotype rh.10 adeno-associated virus (AAV) gene transfer vector expressing the cDNA coding for human FXN; Drug: Prednisone

INTERVENTIONS:
Biological: AAVrh.10hFXN, serotype rh.10 adeno-associated virus (AAV) gene transfer vector expressing the cDNA coding for human FXN — AAVrh.10hFXN will be administered intravenously.
Drug: Prednisone — All participants will remain immunosuppression therapy with prednisone for a total of 14 weeks.

SUMMARY:
The purpose of this study is to test the safety and preliminary efficacy of AAVrh.10hFXN to treat the cardiomyopathy associated with Friedreich's ataxia (FA). AAVrh.10hFXN is a serotype rh.10 adeno-associated virus gene transfer vector coding for Frataxin (FXN). The drug is administered intravenously. This is a phase 1, open label, dose escalation study with a total of 25 participants.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, age 18 to 50
* Willing and able to provide informed consent
* Definitive diagnosis of FA, based on clinical phenotype and genotype (GAA expansion on both alleles)
* >600 GAA repeats in intron 1 in at least one allele
* FARS and SARA neurologic scores consistent with diagnosis of Friedreich's ataxia
* Left ventricle ejection fraction (EF) measured by cardiac MRI of ≥35% to 75%
* Evidence of FA-related cardiac disease, must meet the following criteria: must be abnormal in ≥2 of the following parameters, at least one of which is an abnormal cardiac MRI left ventricular mass index or abnormal cardiopulmonary exercise test

  1. In the absence of other factors known to cause left ventricular hypertrophy, cardiac MRI left ventricular mass index >2 standard deviations above the normal range (males >84 gm/m2, females >69 gm/m2)
  2. Cardiopulmonary arm crank testing with assessment of VO2 max ≤20 mL/kg-min, peak VO2 ≥10 mL/kg-min while maintaining revolutions of ≥40/min. To insure consistency of effort, peak RER ≥1.0
  3. Cardiac MRI stroke volume index <45 mL/m2
  4. Cardiac MRI global longitudinal left ventricular strain <20%
  5. Serum high-sensitivity cardiac troponin above the normal range
* Fibrosis ≤10% in the left ventricular wall on late gadolinium enhancement cardiac MRI
* Resting O2 saturation ≥95%
* Serum neutralizing anti-AAVrh.10 titer <1:125
* Hematocrit >30%
* White blood cell levels within normal limits
* Normal prothrombin, partial thromboplastin time
* Normal liver-related serum parameters (ALT, AST, ALP, bilirubin); normal liver ultrasound and serum alpha fetoprotein
* Normal kidney function as assessed by plasma urea and creatinine; estimated GFR >30 mL/min/1.73m2
* No evidence of active infection of any types, including hepatitis virus (A, B or C), human immunodeficiency virus (HIV-1 and HIV-2), or SARS-CoV2
* Fertile individuals should utilize barrier birth control measures to prevent pregnancy for up to 6 months after vector administration
* Individuals not receiving experimental medications or participating in another experimental protocol for at least 12 wk prior to entry to the study (individuals who are/have received approved therapy will be included).
* Capable of undergoing cardiac MRI
* No contraindications to receiving corticosteroid immunosuppression

Exclusion Criteria:

* Individuals receiving corticosteroids or other immunosuppressive medications
* Individuals with uncontrolled diabetes (glycated hemoglobin, HbA1c levels >7%)
* Genotype FA missense mutation on one or both alleles
* Evidence of infection defined by elevated white blood cell count, temperature >38.5̊ C, infiltrate on chest x-ray
* Decompensated heart failure (NY4A class III-IV at time of baseline clinical assessment)
* Hemoglobin <10 g/dl
* Absolute neutrophil count <1500 cells/mm3
* Platelet count <100,000 cells/mm3
* Hemodynamically unstable atrial or ventricular arrhythmias which require medical intervention
* Contraindication to cardiac MRI (e.g., non-MRI compatible pacemaker/defibrillator) or gadolinium (known or suspected hypersensitivity, glomerular filtration rate <30 mL/min/1.73m2)
* Any malignancy during the last five years, except basal cell skin cancer
* Unrelated clinical condition with life expectancy <12 months (prohibiting follow-up)
* Concomitant conditions (other than FA) known to produce left ventricular hypertrophy, including aortic stenosis, systemic hypertension (BP ≥140/90 on noninvasive blood pressure), or genetically mediated hypertrophic cardiomyopathy
* Use of oxygen supplementation
* Risk for thromboembolic disease, including history of thromboembolic disease hospitalization within the last 90 days, recent trauma and/or recent surgical procedure. If the history of thromboembolic disease is not definitive, the subject will be excluded if laboratory testing suggests a risk for thromboembolic disease because of mutations in the protein-S, protein C, antithrombin, factor V Leiden or prothrombin gene
* Any uncontrolled psychiatric disease
* Pregnant or breastfeeding woman
* Prior participation in any gene and/or cell therapy
* Known obstructive coronary artery disease (as documented by clinical history of myocardial infarction, prior coronary revascularization or angina symptoms (Canadian Cardiovascular Society grade ≥2 at time of baseline clinical assessment), or epicardial obstructive coronary artery disease (≥ 50% left main, ≥ 70% of other major coronary arteries)
* Any lung function abnormalities that would affect cardiopulmonary testing
* Any condition, disorder, or abnormal laboratory test findings at screening which, in the judgment of the investigator, would interfere with the individual's ability to comply with all study requirements, or would require the administration of treatment during the study that could potentially affect the interpretation of the study data, or would place the individual at an unacceptable risk by his/her participation in the study
* If prior infection with SARS-CoV2, any related residual cardiac or pulmonary abnormalities
* Alcoholism or drug addiction (see reference 71 for alcoholism, reference 72 for drug addiction)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-02-22 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety of AAVrh.10hFXN | 5 Years
  To determine the safety of AAVrh.10hFXN, as measured by the number of subjects with any treatment-related adverse events for 5 years.

OTHER OUTCOMES:
Change in cardiopulmonary exercise testing | 5 Years
  To determine changes in parameters of cardiopulmonary testing (measured by the change in VO2max), from screening (pre-treatment) to up to 5 years post administration.
Change in cardiac-relevant parameters in cardiac-magnetic resonance scans | 5 Years
  To determine if there are changes in parameters of cardiac imaging (including Left Ventricular mass, Left Ventricular stroke volume, Global longitudinal strain and wall thickness), from screening (pre-treatment) to up to 5 years post administration.
Change in cardiac-relevant parameters in echocardiograms | 5 Years
  To determine if there are changes in parameters of echocardiograms (including left ventricle mass, Wall thickness and Left ventricle ejection fraction), from screening (pre-treatment) to up to 5 years post administration.
Change in arrhythmias with 24-hour monitoring. | 5 Years
  To determine if there are changes in heart arrhythmias, from screening (pre-treatment) to up to 5 years post administration. This will be measure by holter monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Crystal, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De BP, Cram S, Lee H, Rosenberg JB, Sondhi D, Crystal RG, Kaminsky SM. Assessment of Residual Full-Length SV40 Large T Antigen in Clinical-Grade Adeno-Associated Virus Vectors Produced in 293T Cells. Hum Gene Ther. 2023 Aug;34(15-16):697-704. doi: 10.1089/hum.2023.032. PMID 37171121